CLINICAL TRIAL: NCT04945122
Title: Comparison of Atorvastatin and Pitavastatin on the Effect of HbA1c in Acute Myocardial Infarction (AMI) Patients With Abnormal Glucose Metabolism: a Multicenter Prospective Randomized Clinical Trial
Brief Title: Comparison of Atorvastatin and Pitavastatin on the Effect of HbA1c in AMI Patients With Abnormal Glucose Metabolism
Acronym: CAPE-AMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Yuejin Yang, Vice President of Fuwai Hospital, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-685
Record Dates: First submitted 2018-01-23; First posted 2021-06-30 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Acute Myocardial Infarction; Glucose Metabolism Disorders
Keywords: Pitavastatin; Atorvastatin; HbA1c; LDL-C
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — pitavastatin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pitavastatin (Experimental): Patients diagnosed AMI with abnormal glucose metabolism use pitavastatin (4mg po Qn) to control cholesterol for 6 months.
  Interventions: Drug: Pitavastatin
- Atorvastatin (Active Comparator): Patients diagnosed AMI with abnormal glucose metabolism use atorvastatin (20mg po Qn) to control cholesterol for 6 months.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Pitavastatin — Pitavastatin 4mg Qn
  Arms: Pitavastatin
Drug: Atorvastatin — Atorvastatin 20mg Qn
  Other Names: Lipitor
  Arms: Atorvastatin

SUMMARY:
Different types of statins show different influences on glycometabolism. There are no systemic analyses of the effects that statins exert on the metabolism of glucoses so far in China. This research aims to compare impacts on the glycometabolism of pitavastatin in AMI patients with atorvastatin and to accumulate data for guiding the utilization of statins.

DETAILED DESCRIPTION:
General study design:

This study is a prospective, multicenter, open and randomized controlled clinical trial, which utilize online registration database of CAMI to do the enrollment, randomization and follow-up. We will select 14 of the centers to compete into the group. The researchers used a central randomized distribution system to prescribe medication for patients. Follow the method of drug administration approved by the state drug administration department, we will estimate the efficacy and safety of treatment at the following timing: baseline, one month and six months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed acute myocardial infarction.
2. Diabetes or pre-diabetes.
3. The patient signed informed consent.

Exclusion Criteria:

1. A clear history of chronic liver disease, or abnormal liver function (ALT/AST>1.5×ULN).
2. There is evidence of active inflammatory myopathy or CK>3×ULN.
3. Being allergic to statins or severe side effects were caused by taking statins(including myolysis).
4. Combined with hypothyroidism, nephrotic syndrome, alcoholism, pancreatitis, lupus erythematosus.
5. All patients who had a clear adverse reaction to the statins.
6. Possibility of pregnancy, pregnant or lactating patients.
7. There may be limited medical history of subjects who may can not complete their treatment during the study period.
8. Undergoing or planning to functional renal transplantation.
9. The life expectancy is no more than half a year.
10. Patients who are taking birth control pills, steroid hormones and imidazole drugs.
11. Patients who have participated in clinical trials of other drugs within 1 month, or known that clinical follow-up or research on drug compliance poorly.
12. Patients are not fit to be tested according to the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c reduction | six months after treatment
  Comparing the impact on HbA1c of AMI patients with abnormal glucose metabolism using pitavastatin 4mg versus atorvastatin 20mg

SECONDARY OUTCOMES:
LDL-c reduction | six months after treatment
  Comparing the absolute reduction of LDL-c level in AMI patients with abnormal glucose metabolism using pitavastatin 4mg versus atorvastatin 20mg

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-jin Gao, M.D., Principal Investigator — National Center for Cardiovascular Diseases, CAMS and Peking Union Medical College, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoy SM. Pitavastatin: A Review in Hypercholesterolemia. Am J Cardiovasc Drugs. 2017 Apr;17(2):157-168. doi: 10.1007/s40256-017-0213-8. PMID 28130659
- [Background] Yoon D, Sheen SS, Lee S, Choi YJ, Park RW, Lim HS. Statins and risk for new-onset diabetes mellitus: A real-world cohort study using a clinical research database. Medicine (Baltimore). 2016 Nov;95(46):e5429. doi: 10.1097/MD.0000000000005429. PMID 27861386
- [Background] China Cholesterol Education Program (CCEP) Working Committee; Atherosclerosis Thrombosis Prevention and Control Subcommittee of Chinese International Exchange and Promotion Association for Medical and Healthcare; Cardiovascular Disease Subcommittee of China Association of Gerontology and Geriatrics; Atherosclerosis Professional Committee of Chinese College of Cardiovascular Physicians. [China cholesterol education program (CCEP) expert advice for the management of dyslipidaemias to reduce cardiovascular risk (2019)]. Zhonghua Nei Ke Za Zhi. 2020 Jan 1;59(1):18-22. doi: 10.3760/cma.j.issn.0578-1426.2020.01.003. Chinese. PMID 31887831
- [Background] Livingstone SJ, Looker HC, Akbar T, Betteridge DJ, Durrington PN, Hitman GA, Neil HA, Fuller JH, Colhoun HM. Effect of atorvastatin on glycaemia progression in patients with diabetes: an analysis from the Collaborative Atorvastatin in Diabetes Trial (CARDS). Diabetologia. 2016 Feb;59(2):299-306. doi: 10.1007/s00125-015-3802-6. Epub 2015 Nov 17. PMID 26577796
- [Background] Huang CH, Huang YY, Hsu BR. Pitavastatin improves glycated hemoglobin in patients with poorly controlled type 2 diabetes. J Diabetes Investig. 2016 Sep;7(5):769-76. doi: 10.1111/jdi.12483. Epub 2016 Feb 22. PMID 27181110
- [Background] Nakagomi A, Shibui T, Kohashi K, Kosugi M, Kusama Y, Atarashi H, Shimizu W. Differential Effects of Atorvastatin and Pitavastatin on Inflammation, Insulin Resistance, and the Carotid Intima-Media Thickness in Patients with Dyslipidemia. J Atheroscler Thromb. 2015;22(11):1158-71. doi: 10.5551/jat.29520. Epub 2015 Jun 17. PMID 26084792
- [Background] Choi SH, Lim S, Hong ES, Seo JA, Park CY, Noh JH, Mok JO, Lee KY, Park JS, Kim DJ, Lee CB, Kim SR, Jang HC. PROPIT: A PROspective comparative clinical study evaluating the efficacy and safety of PITavastatin in patients with metabolic syndrome. Clin Endocrinol (Oxf). 2015 May;82(5):670-7. doi: 10.1111/cen.12580. Epub 2014 Oct 17. PMID 25109606
- [Background] Cho Y, Choe E, Lee YH, Seo JW, Choi Y, Yun Y, Wang HJ, Ahn CW, Cha BS, Lee HC, Kang ES. Risk of diabetes in patients treated with HMG-CoA reductase inhibitors. Metabolism. 2015 Apr;64(4):482-8. doi: 10.1016/j.metabol.2014.09.008. Epub 2014 Sep 28. PMID 25312577
- [Background] Baudrand R, Pojoga LH, Vaidya A, Garza AE, Vohringer PA, Jeunemaitre X, Hopkins PN, Yao TM, Williams J, Adler GK, Williams GH. Statin Use and Adrenal Aldosterone Production in Hypertensive and Diabetic Subjects. Circulation. 2015 Nov 10;132(19):1825-33. doi: 10.1161/CIRCULATIONAHA.115.016759. Epub 2015 Oct 2. PMID 26432671
- [Background] Arnaboldi L, Corsini A. Could changes in adiponectin drive the effect of statins on the risk of new-onset diabetes? The case of pitavastatin. Atheroscler Suppl. 2015 Jan;16:1-27. doi: 10.1016/S1567-5688(14)70002-9. PMID 25575403
- [Background] Sponseller CA, Morgan RE, Kryzhanovski VA, Campbell SE, Davidson MH. Comparison of the lipid-lowering effects of pitavastatin 4 mg versus pravastatin 40 mg in adults with primary hyperlipidemia or mixed (combined) dyslipidemia: a Phase IV, prospective, US, multicenter, randomized, double-blind, superiority trial. Clin Ther. 2014 Aug 1;36(8):1211-22. doi: 10.1016/j.clinthera.2014.06.009. Epub 2014 Jul 3. PMID 24998014
- [Background] Navarese EP, Buffon A, Andreotti F, Kozinski M, Welton N, Fabiszak T, Caputo S, Grzesk G, Kubica A, Swiatkiewicz I, Sukiennik A, Kelm M, De Servi S, Kubica J. Meta-analysis of impact of different types and doses of statins on new-onset diabetes mellitus. Am J Cardiol. 2013 Apr 15;111(8):1123-30. doi: 10.1016/j.amjcard.2012.12.037. Epub 2013 Jan 24. PMID 23352266
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Warita S, Kawasaki M, Tanaka R, Ono K, Kojima T, Hirose T, Iwama M, Watanabe T, Nishigaki K, Takemura G, Noda T, Watanabe S, Minatoguchi S. Effects of pitavastatin on cardiac structure and function and on prevention of atrial fibrillation in elderly hypertensive patients: a prospective study of 2-years' follow-up. Circ J. 2012;76(12):2755-62. doi: 10.1253/circj.cj-12-0722. Epub 2012 Aug 8. PMID 22878405
- [Background] Yokote K, Shimano H, Urashima M, Teramoto T. Efficacy and safety of pitavastatin in Japanese patients with hypercholesterolemia: LIVES study and subanalysis. Expert Rev Cardiovasc Ther. 2011 May;9(5):555-62. doi: 10.1586/erc.11.47. PMID 21615316
- [Background] Preiss D, Seshasai SR, Welsh P, Murphy SA, Ho JE, Waters DD, DeMicco DA, Barter P, Cannon CP, Sabatine MS, Braunwald E, Kastelein JJ, de Lemos JA, Blazing MA, Pedersen TR, Tikkanen MJ, Sattar N, Ray KK. Risk of incident diabetes with intensive-dose compared with moderate-dose statin therapy: a meta-analysis. JAMA. 2011 Jun 22;305(24):2556-64. doi: 10.1001/jama.2011.860. PMID 21693744
- [Background] Gumprecht J, Gosho M, Budinski D, Hounslow N. Comparative long-term efficacy and tolerability of pitavastatin 4 mg and atorvastatin 20-40 mg in patients with type 2 diabetes mellitus and combined (mixed) dyslipidaemia. Diabetes Obes Metab. 2011 Nov;13(11):1047-55. doi: 10.1111/j.1463-1326.2011.01477.x. PMID 21812889
- [Background] Yoshika M, Komiyama Y, Masuda M, Yokoi T, Masaki H, Ohkura H, Takahashi H. Pitavastatin further decreases serum high-sensitive C-reactive protein levels in hypertensive patients with hypercholesterolemia treated with angiotensin II, type-1 receptor antagonists. Clin Exp Hypertens. 2010;32(6):341-6. doi: 10.3109/10641961003628460. PMID 21028996
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Ridker PM, Macfadyen JG, Nordestgaard BG, Koenig W, Kastelein JJ, Genest J, Glynn RJ. Rosuvastatin for primary prevention among individuals with elevated high-sensitivity c-reactive protein and 5% to 10% and 10% to 20% 10-year risk. Implications of the Justification for Use of Statins in Prevention: an Intervention Trial Evaluating Rosuvastatin (JUPITER) trial for "intermediate risk". Circ Cardiovasc Qual Outcomes. 2010 Sep;3(5):447-52. doi: 10.1161/CIRCOUTCOMES.110.938118. Epub 2010 Aug 24. PMID 20736443
- [Background] Yamakawa T, Takano T, Tanaka S, Kadonosono K, Terauchi Y. Influence of pitavastatin on glucose tolerance in patients with type 2 diabetes mellitus. J Atheroscler Thromb. 2008 Oct;15(5):269-75. doi: 10.5551/jat.e562. PMID 18981652
- [Background] Ridker PM, Danielson E, Fonseca FA, Genest J, Gotto AM Jr, Kastelein JJ, Koenig W, Libby P, Lorenzatti AJ, MacFadyen JG, Nordestgaard BG, Shepherd J, Willerson JT, Glynn RJ; JUPITER Study Group. Rosuvastatin to prevent vascular events in men and women with elevated C-reactive protein. N Engl J Med. 2008 Nov 20;359(21):2195-207. doi: 10.1056/NEJMoa0807646. Epub 2008 Nov 9. PMID 18997196